CLINICAL TRIAL: NCT01650623
Title: Gait Training Associated With Executive Functions Tasks in Subjects With Parkinson´s Disease: A Randomised Controlled Trial
Brief Title: Gait Training With Executive Functions Tasks in Subjects With Parkinson´s Disease: A Randomised Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Coordination for the Improvement of Higher Education Personnel (Other)
Responsible Party: Principal Investigator, Cynthia Bedeschi Ferrari, PT, Ms, PhD Student - Neuroscience and Behavior, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USPNEC002
Record Dates: First submitted 2012-07-19; First posted 2012-07-26 (Estimated); Last update posted 2012-11-08 (Estimated); Status verified 2012-11

CONDITIONS: Parkinson´s Disease
Keywords: Parkinson´s Disease; Rehabilitation; Cognition
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gait training executive functions tasks (Experimental): The experimental group will perform a gait training associated with the tasks that require the main executive functions (dual-task condition).
  Interventions: Behavioral: Gait training executive functions tasks
- Gait training alone (Active Comparator): The control group will perform a gait training alone, without associated tasks (single-task condition).
  Interventions: Behavioral: Gait training alone

INTERVENTIONS:
Behavioral: Gait training executive functions tasks — The training will consist of 10 sessions, two times per week for five weeks, and consists of 30 minutes of global exercises that involves stretching, muscle strengthen and axial mobility exercises, and another 30 minutes of gait training in a dual-task condition associated with distracting tasks that require handling of the main executive functions: volition, self-awareness, planning, response inhibition, response monitoring and attention.
  Arms: Gait training executive functions tasks
Behavioral: Gait training alone — The training will consist of 10 sessions, two times per week for five weeks, and consists of 30 minutes of global exercises that involves stretching, muscle strengthen and axial mobility exercises, and another 30 minutes of gait training alone, without other tasks.
  Arms: Gait training alone

SUMMARY:
The aim of this study is to compare two physical therapy training consisting of gait training that are distinguished by one being associated with tasks that require handling of the main executive functions, performed by individuals with Parkinson's Disease.

The investigators hypothesis is that the experimental group (EG), which hold gait training with higher cognitive demands (dual-task condition), will make improvements in the parameters measured (functionality of gait and cognitive ability) to a greater extent compared to the control group (CG), which hold gait training without executive tasks (single-task condition).

DETAILED DESCRIPTION:
The aim of this study is to compare two physical therapy training consisting of a gait training that are distinguished by one being associated with tasks that require handling of the main executive functions (protocol designed by the same team), performed by individuals with Parkinson's Disease.

Both training consists of 30 minutes of global exercises that involves stretching, muscle strengthen and axial mobility exercises, with the following difference:

* the experimental group (EG) will hold another 30 minutes of gait training in a dual-task condition associated with distracting tasks that require handling of the main executive functions;
* the control group (CG) will hold an additional 30 minutes of gait training without associated tasks.

It will be a prospective study, single blind, randomized, where 30 patients with PD in stages 1 to 3 on Hoehn & Yahr scale will participate in the study, to be held in Brazil Parkinson Association. Patients will be randomized into an experimental and control group, 15 in each one.

The training will consist of 10 sessions, two times per week for five weeks. The executive tasks concomitant with gait training cover the following executive functions: volition, self-awareness, planning, response inhibition, response monitoring and attention.

The main outcome measures are: (1) Dynamic Gait Index (DGI), (2) Montreal Cognitive Assessment (MoCA), (3) Trail Making Test A and B, (4) Unified Parkinson's Disease Rating Scale (UPDRS) and (5) Falls Efficacy Scale (FES).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Idiopathic PD performed by a neurologist specialist in movement disorders;
* In use of dopaminergic medication;
* Disease severity of 1 to 3 according to Hoehn & Yahr scale;
* Absence of other neurological disorders or co-morbidities that may affect gait;
* Absence of dementia (score above 24 on the Mini Mental State Examination - MMSE);
* Vision and hearing adequate or corrected to normal;
* Ability to walk independently;
* Absence of prolonged off state;
* Age 50 to 85 years.

Exclusion Criteria:

* Biomechanical alterations (other pathologies) that could compromise the completion of training;
* Presence of depression, detected by the Geriatric Depression Scale (GDS-15);
* Presence of any neurological, auditory or visual deficit that could compromise distracting task performance during gait training;
* Any changes in drug treatment for PD.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-05 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Dynamic Gait Index | 05/2013 (Up to ten months)
  The scale assesses the ability to adapt the gait during motor tasks with different demands.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | 05/2013 (Up to ten months)
  This scale was developed in order to detect mild degrees of cognitive impairment. The instrument assesses different cognitive domains such as attention and concentration, executive functions, memory, language, visuo-constructive skills, calculations, and orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elisa P Piemonte, PhD, Study Director — University of Sao Paulo; Cynthia B Ferrari, PhD Student, Principal Investigator — University of Sao Paulo
Locations (1):
- Brazil Parkinson Association, São Paulo, São Paulo, Brazil